CLINICAL TRIAL: NCT02533193
Title: A Randomized Controlled Trial of Enhanced Recovery After Surgery Protocal Versus Traditional Care in Laparoscopic Hepatectomy
Brief Title: Enhanced Recovery After Surgery Protocal Versus Traditional Care in Laparoscopic Hepatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Xiujun Cai, President, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sirrrsh20150802-1
Record Dates: First submitted 2015-08-11; First posted 2015-08-26 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Liver Diseases
Keywords: enhanced recovery after surgery protocal; laparoscopic hepatectomy
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- enhanced recovery after surgery protocal (Active Comparator): ERAS perioperative cares patients planned to undergoing laparoscopic gastrectomy, following the ERAS protocols.
  Interventions: Procedure: ERAS perioperative cares
- Conventional perioperative cares (Active Comparator): Conventional perioperative cares patents will be managed by our hospital's critical pathways.
  Interventions: Procedure: Conventional perioperative cares

INTERVENTIONS:
Procedure: ERAS perioperative cares — 1. Patient's preoperative counseling & education before surgery
  2. No Bowel preparation
  3. Drug: Oral Carbohydrate Solution (OCS). Take 250ml OCS orally 2 hours before surgery
  4. Fluid restriction & Management by pulse contour analysis or transesophageal doppler
  5. Early mobilization
  6. Early oral feeding (postoperative 1 day - liquid diet, 2 days - semifluid diet (SFD), 3 days - normal diet)
  7. Intravenous patient controlled analgesics (no opioids analgesics)
  8. Postoperative Nausea Active Control
  9. No nasogastric tube
  10. No drain insertion
  11. Patients will be discharged at POD#4 if there's no problem
  Arms: enhanced recovery after surgery protocal
Procedure: Conventional perioperative cares — 1. No Patient's preoperative counseling & education before surgery
  2. Bowel preparation
  3. No Oral Carbohydrate Solution (OCS) loading until 2hours before surgery
  4. Conventional Fluid Management by clinical signs (Urine output, heart rate etc.)
  5. Conventional Mobilization
  6. Conventional oral feeding (POD#2 SOW, #3 SFD, #4 SBD)
  7. IV PCA
  8. Postoperative Nausea Control if needed
  9. No Thromboembolism prophylaxis
  10. No or Low Content Oxygen therapy
  11. Drainage tube insertion if needed
  Arms: Conventional perioperative cares

SUMMARY:
The purpose of this study is to investigate the clinical value of enhanced recovery after surgery protocal in laparoscopic hepatectomy by assessing its outcomes and hospital stay days comparing with traditional care .

DETAILED DESCRIPTION:
The ERAS programs has been proved to be a useful solutions in patients undergoing colorectal surgery in terms of significantly reduced postoperative complications and shorter length of hospital stay, compared to the patients of conventional treatment.

But few studies reported about the ERAS programs in the laparoscopic hepatectomy.

The purpose of this study is to investigate the clinical value of enhanced recovery after surgery protocal in laparoscopic hepatectomy by assessing its outcomes and hospital stay days comparing with traditional care .

ELIGIBILITY:
Inclusion Criteria:

* If patients were diagnosed with tumors

  1. Located at segment Ⅱ、Ⅲ、Ⅳb、Ⅴ or Ⅵ
  2. The tumor location and size do not affect the dissection of hepatic hilar region
  3. Tumor size less than 10cm
  4. Without portal vein tumor thrombus
  5. Without intrahepatic or distant metastasis
* Partial resection or half liver resection
* Willingness to participate in the study
* Able to understand the nature of the study and what will be required of them
* Body mass index of between 18 and 35
* Child-Pugh classification of A to B
* American Society of Anesthesiologists (ASA) grading of I to III

Exclusion Criteria:

* Pregnant or lactating women
* Unwillingness to participate
* Inability to give written informed consent
* Child-Pugh classification of C
* ASA grading of IV to V
* Tumor invasion of the inferior vena cava or confluence part of hepatic vein
* Decompensated liver cirrhosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
post-operative hospital stay | up to 4 weeks after surgery
  participants will be followed for the duration of hospital stay, an expected average of 6 days
Recovering Rate | 6 days after surgery
  1. No major complication
  2. Tolerance of semiliquid diet
  3. Normal activity
  4. Good pain control with analgesic-free or oral analgesics.

SECONDARY OUTCOMES:
Time to functional recovery (days from operation to functional recovery) | up to 4 weeks after surgery
  Normal or decreasing serum bilirubin Good pain control with oral analgesia only Tolerance of solid food No intravenous fluids Mobile independently or at the preoperative level All of the above is functional recovery.
cost of hospitalization | up to 1 month after surgery
  medical expense
Quality of life | up to 1 month after surgery
  EQ-5d health questionnaire and Kolcaba's GCQ (General Comfort Questionnaire), before the operation, on postoperation 1 day, postoperation 3 day, postoperation 5 day, postoperation 1 month
operation time | the day of surgery
associated cytokines in peripheral blood (IL-6, IL-10 and TNF-α) | before the operation, on postoperation 1 day, postoperation 2 day, postoperation 4 day
  associated cytokines in peripheral blood were tested on preoperation, postoperation Day1, postoperation Day2, postoperation Day4
liver function | up to 1 month after surgery
  liver function were tested on preoperation, postoperation Day1, postoperation Day2, postoperation Day4, postoperation 1 month if PT ≥ 50% and TB ≥ 50 μmol/L， it supports the liver dysfunction.
Visual Analog Score for pain | up to 5 days after surgery
  postoperative 2hours, 6 hours, 1 days, 2 days, 3 days, 4 days and 5 days
Estimated blood loss | the day of surgery
  blood loss during the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Institute of Minimally Invasive Surgery, Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China